CLINICAL TRIAL: NCT05575388
Title: Pattern of Isolated Fungi From Bronchoalveolar Lavage Among Patients With Lung Cancer, a Prospective Cross Sectional Study.
Brief Title: Pattern of Isolated Fungi From Bronchoalveolar Lavage Among Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MS/353
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer
Keywords: lung cancer, fungal colonization, fiberoptic bronchoscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the prevalence and pattern of isolated fungi from patients with lung cancer at the time of diagnosis.

DETAILED DESCRIPTION:
The role of infection as a cause of lung cancer is still being debated. Also, identification of potentially pathogenic organisms colonizing the lower respiratory tract in patients with lung cancer is important as this may increase the risk of lung infections in the natural course of lung cancer that can restrain the effect of oncological treatment and affect their survival (Klastersky and Aoun, 2004). Screening those cases for fungal colonization of the respiratory tract would characterize patients who needed closer monitoring for the occurrence of potential complications such as acute invasive fungal infection (Biswas et al., 2010).

Aim of the study The aim of the study is to detect the prevalence and pattern of isolated fungi from patients with lung cancer at the time of diagnosis before starting chemotherapy or radiotherapy.

Patients:

Inclusion criteria:

Patients presented to chest medicine department outpatient clinic with radiological and/or clinical manifestations suspicious of lung cancer such as a hilar mass, collapse or unresolved consolidation with accompanying volume loss according to Hollings and Shawn, (2000), will be subjected to FOB for diagnosis. Those definitely diagnosed as central bronchogenic carcinoma will be included in the study.

Exclusion criteria:

* Patients with active tuberculosis.
* Patients with HIV (human immunodeficiency virus) infection.
* Presence of neutropenia defined as an absolute neutrophil count (ANC) < 1,000/µL (equivalent to < 1.0 × 109/L) according to Taplitz et al., (2018).
* Patients on systemic corticosteroids therapy.
* Patients on chemotherapy or radiotherapy.
* Patients on antifungal therapy.
* Patients with absolute contraindications to FOB including who were hemodynamically unstable or with platelet counts could not be maintained over 50 × 109 /l or INR > 1.5 and patients with refractory hypoxemia.

Study design:

This is cross-sectional prospective study

Methods:

All patients will be subjected to the following:

1. Demographic data (age and sex), smoking history and co-morbid diseases as COPD, hypertension (HTN), diabetes mellitus (DM), ischemic heart disease, bronchial asthma (BA) and previous malignancy.
2. Full history taking with stress on dyspnea, cough, chest pain, hemoptysis, toxemic symptoms and compressive manifestations.

   1. Dyspnea score was evaluated according to The MRC breathlessness scale (2008).
   2. Hemoptysis score was evaluated according to the amount of blood expectorated in 24 h into as mild (< 30 ml), moderate (31-100 ml), severe (100-600 ml) and massive (> 600 mL) according to Ozgül et al., (2005).
   3. Cough score assessment from 0 to 5 according to Hsu et al., (1994).
   4. Chest pain scoring was done according to The McGill Pain Questionnaire (Melzack, 1987).
3. General and local chest examination.
4. Laboratory work up:

   1. Complete blood count(CBC).
   2. Liver function tests.
   3. Serum creatinine.
   4. Coagulation profile (prothrombin time, INR, APTT and platelet count).
   5. Virology profile (HBV, HCV and HIV).
5. Radiological assessment (Chest X-ray and CT chest):

   1. Description either nodule, mass, cavity, consolidation or ground glass opacity according to Hollings and Shawn, (2000).
   2. Evaluation of the tumor size ,site of and its effect on lobar or total lung collapse.
   3. Hilar and mediastinal lymphadenopathy assessment according to El-Sherief et al., (2004).
   4. Presence of pleural effusion.
   5. Chest wall invasion.

Bronchoscopic procedures FOB examination will be performed using the video-bronchoscopes (PENTAX EB 1575 K) manufactured by Pentax Company Tokyo, Japan.

Bronchoscopic findings will be interpretated into:

1. Visible tumors may be either:

   1. Tumor protruding from the bronchial wall into the bronchial lumen.
   2. Nodular mucosa without definitive mass.
2. Bronchial wall distortion: the mucosa appears normal but there are secondary effects produced by tumor such as compression, edema or stenosis.
3. No abnormality detected.

Preservation of samples:

1. The BAL fluid will be collected in two sterile containers and transported immediately, one sample to the mycology laboratory and the other to cytological lab.
2. Tissue samples will be divided into 2 parts:

   1. Part (A) will be put in saline containing tube that will be transferred to the microbiology laboratory for staining for fungi and fungus culture.
   2. Part (B) will be preserved in formalin 10% for histopathological examination of the tumor, cell typing with Hematoxylin and Eosin and immunostaining when needed as well as staining for fungi in lung tumor biopsies with silver stain .

Diagnostic criteria for fungal infection will be considered according to De Pauw et al., (2008):

Proven" fungal infection : positive fungal culture or histological demonstration of fungal or hyphal elements in a specimen of the diseased tissue excluding bronchoalveolar lavage.

Fungus colonization : positive fungal culture in patients who do not meet the above criteria for proven .

ELIGIBILITY:
Inclusion criteria

* All patients definitely diagnosed as central bronchogenic carcinoma from positive cytopathology of specimens taken through investigation by FOB before receiving any specific treatment.

Exclusion criteria:

* the presence of neutropenia with an absolute neutrophil count < 1,000/µL (equivalent to < 1.0 × 109/L)
* patients on systemic corticosteroids therapy or those on chemotherapy or radiotherapy or antifungal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients definitely diagnosed as central bronchogenic carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
number of participants with positive fungal growth | April 2018 and October 2020
  assessed by fungal culture of BAL

SECONDARY OUTCOMES:
predictors of fungal infection in lung cancer participants | April 2018 and October 2020
  assessed by comparing lung cancer cases with fungal infection vs those with negative fungal growth as regards characteristics of the participants and cell types of lung cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Al Mansurah, Egypt